CLINICAL TRIAL: NCT05420649
Title: Evaluation of the Feasibility and Safety of Laryngoscopic Microsurgery Under Non-intubation Anesthesia With Combination of Superior Laryngeal Nerve Block
Brief Title: Evaluation of the Feasibility and Safety of Laryngoscopic Microsurgery Under Non-intubation Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Yuan-Yi Chia, Chief of Anesthesiology, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KSVGH20-CT9-09
Record Dates: First submitted 2022-05-03; First posted 2022-06-15 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Spontaneous Breathing; Laryngomicrosurgery; Superior Laryngeal Nerve Block
Keywords: Nonintubated; Spontaneous breathing; Laryngomicrosurgery; Superior laryngeal nerve block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intubated general anesthesia LMS (No Intervention): Patients received LMS with intubated general anesthesia
- Non-intubated LMS with apnea (Experimental): Patients received non-intubated LMS with administration of muscle relaxant and optiflow(HFNO) device.
  Interventions: Procedure: Non-intubated Laryngomicrosurgery
- Non-intubated LMS with spontaneous breathing (Experimental): Patients received non-intubated LMS optiflow(HFNO) device and maintained spontaneous breathing.
  Interventions: Procedure: Non-intubated Laryngomicrosurgery

INTERVENTIONS:
Procedure: Non-intubated Laryngomicrosurgery — Non-intubated LMS was performed with assistance of Optiflow (HFNO).
  Arms: Non-intubated LMS with apnea; Non-intubated LMS with spontaneous breathing

SUMMARY:
Nonintubated anesthesia applied in combination with high-flow nasal oxygen (HFNO) is an alternative strategy for laryngeal microsurgery (LMS). LMS is a common procedure in otolaryngology that typically requires endotracheal tube intubation under general anesthesia. Endotracheal tube intubation causes complications; a nonintubated strategy can avoid these complications and provide a clearer surgical field of vision, enabling vocal cord inspection and disposal. Administering a muscle relaxant can also help prevent bucking during surgery but can engender apnea and hypercapnia, which may have negative effects on hemodynamics. Therefore, the investigators assessed the effectiveness of a superior laryngeal nerve block (SLNB) with intravenous general anesthesia in maintaining spontaneous breathing and improving safety during LMS with nonintubated anesthesia.

DETAILED DESCRIPTION:
Laryngeal microsurgery (LMS) is among the most common operations in otolaryngology and typically requires general anesthesia administered through endotracheal tube intubation. Endotracheal tube intubation provides stable gas exchange, protects the airways by preventing secretions from falling into the lower respiratory tract, and enables the monitoring of parameters such as tidal volume and end-tidal CO2.

Nonintubated anesthesia applied in combination with transnasal humidified rapid-insufflation ventilatory exchange or high-flow nasal oxygen (HFNO) is another option for LMS. LMS with nonintubated anesthesia can avoid the complications caused by endotracheal tube intubation such as oral tissue trauma, tracheal trauma, and dental injury. Furthermore, LMS with nonintubated anesthesia can provide a clearer surgical field of vision that allows the vocal cords to be inspected and disposed of completely. Current practice in LMS with nonintubated anesthesia is to administer a muscle relaxant to help avoid bucking during the procedure. However, the administration of a muscle relaxant can lead to apnea and hypercapnia, which may negatively affect hemodynamics. Therefore, the investigators investigated the use of a superior laryngeal nerve block (SLNB) with intravenous general anesthesia to help the patient maintain spontaneous breathing and provide higher surgical safety during LMS with nonintubated anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* The patient who needed to undergo LMS.

Exclusion Criteria:

* Severe airway obstruction.
* Severe airway disease.
* American Society of anesthesiologists (ASA) physical state > III.
* Pregnancy or body mass index (BMI) ≥ 40 kg/m2.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
PaCO2 after Laryngomicrosurgery | ABG was measured immediately after the end of LMS
  ABG was measured immediately after the end of LMS

SECONDARY OUTCOMES:
pH after Laryngomicrosurgery | ABG was measured immediately after the end of LMS
  ABG was measured immediately after the end of LMS
Heart rate (HR) | during the LMS procedure
  Hemodynamic data were measured every 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Yi Chia, Director, Principal Investigator — Kaohsiung Veterans General Hospital.; Yu Ting Kuo, physician, Study Director — Kaohsiung Veterans General Hospital.; Ting Shou Chang, physician, Study Director — Kaohsiung Veterans General Hospital.; Chih Chi Tsai, RA, Study Chair — Kaohsiung Veterans General Hospital.; Li-Ya Tseng, physician, Study Director — Kaohsiung Veterans General Hospital.; Pei-Wen Shen, physician, Study Director — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Booth AWG, Vidhani K, Lee PK, Thomsett CM. SponTaneous Respiration using IntraVEnous anaesthesia and Hi-flow nasal oxygen (STRIVE Hi) maintains oxygenation and airway patency during management of the obstructed airway: an observational study. Br J Anaesth. 2017 Mar 1;118(3):444-451. doi: 10.1093/bja/aew468. PMID 28203745
- [Background] Montgomery J, Melia L, O'Donnell N, MacKenzie K. Intubation trauma and the head and neck surgeon: issues with a shared airway. J R Soc Med. 2015 Nov;108(11):426-8. doi: 10.1177/0141076815614803. No abstract available. PMID 26609095
- [Background] Yang SH, Wu CY, Tseng WH, Cherng WY, Hsiao TY, Cheng YJ, Chan KC. Nonintubated laryngomicrosurgery with Transnasal Humidified Rapid-Insufflation Ventilatory Exchange: A case series. J Formos Med Assoc. 2019 Jul;118(7):1138-1143. doi: 10.1016/j.jfma.2018.11.009. Epub 2018 Dec 3. PMID 30522856
- [Background] Catalano G, Robeel RA, Cheney GA, Spurling BC, Catalano MC, Schultz SK, Sanchez DL. Antidepressant Augmentation: A Review of the Literature and a Review of the Pharmacoeconomic Considerations. J Clin Psychopharmacol. 2020 Jul/Aug;40(4):396-400. doi: 10.1097/JCP.0000000000001236. PMID 32639292
- [Background] Yasar NF, Uylas MU, Badak B, Bilge U, Oner S, Ihtiyar E, Caga T, Pasaoglu E. Can we predict mortality in patients with necrotizing fasciitis using conventional scoring systems? Ulus Travma Acil Cerrahi Derg. 2017 Sep;23(5):383-388. doi: 10.5505/tjtes.2016.19940. PMID 29052823
- [Background] Booth AWG, Vidhani K, Lee PK, Coman SH, Pelecanos AM, Dimeski G, Sturgess DJ. The Effect of High-Flow Nasal Oxygen on Carbon Dioxide Accumulation in Apneic or Spontaneously Breathing Adults During Airway Surgery: A Randomized-Controlled Trial. Anesth Analg. 2021 Jul 1;133(1):133-141. doi: 10.1213/ANE.0000000000005002. PMID 32618626
- [Background] Parke RL, Bloch A, McGuinness SP. Effect of Very-High-Flow Nasal Therapy on Airway Pressure and End-Expiratory Lung Impedance in Healthy Volunteers. Respir Care. 2015 Oct;60(10):1397-403. doi: 10.4187/respcare.04028. Epub 2015 Sep 1. PMID 26329355
- [Background] Williams R, Rankin N, Smith T, Galler D, Seakins P. Relationship between the humidity and temperature of inspired gas and the function of the airway mucosa. Crit Care Med. 1996 Nov;24(11):1920-9. doi: 10.1097/00003246-199611000-00025. PMID 8917046
- [Background] Bernards CM, Knowlton SL, Schmidt DF, DePaso WJ, Lee MK, McDonald SB, Bains OS. Respiratory and sleep effects of remifentanil in volunteers with moderate obstructive sleep apnea. Anesthesiology. 2009 Jan;110(1):41-9. doi: 10.1097/ALN.0b013e318190b501. PMID 19104169
- [Background] Stockwell M, Lozanoff S, Lang SA, Nyssen J. Superior laryngeal nerve block: an anatomical study. Clin Anat. 1995;8(2):89-95. doi: 10.1002/ca.980080202. PMID 7712327
- [Background] Manikandan S, Neema PK, Rathod RC. Ultrasound-guided bilateral superior laryngeal nerve block to aid awake endotracheal intubation in a patient with cervical spine disease for emergency surgery. Anaesth Intensive Care. 2010 Sep;38(5):946-8. doi: 10.1177/0310057X1003800523. PMID 20865885
- [Background] Pani N, Kumar Rath S. Regional & topical anaesthesia of upper airways. Indian J Anaesth. 2009 Dec;53(6):641-8. PMID 20640090
- [Background] Menda F, Koner O, Sayin M, Ture H, Imer P, Aykac B. Dexmedetomidine as an adjunct to anesthetic induction to attenuate hemodynamic response to endotracheal intubation in patients undergoing fast-track CABG. Ann Card Anaesth. 2010 Jan-Apr;13(1):16-21. doi: 10.4103/0971-9784.58829. PMID 20075530
- [Background] Chopra P, Dixit MB, Dang A, Gupta V. Dexmedetomidine provides optimum conditions during awake fiberoptic intubation in simulated cervical spine injury patients. J Anaesthesiol Clin Pharmacol. 2016 Jan-Mar;32(1):54-8. doi: 10.4103/0970-9185.175666. PMID 27006542
- [Background] Michard F. Changes in arterial pressure during mechanical ventilation. Anesthesiology. 2005 Aug;103(2):419-28; quiz 449-5. doi: 10.1097/00000542-200508000-00026. PMID 16052125
- [Background] Funk DJ. Apneic oxygenation: Let's all just take a deep breath. Can J Anaesth. 2017 Apr;64(4):358-360. doi: 10.1007/s12630-016-0801-0. Epub 2016 Dec 22. No abstract available. PMID 28008564
- [Background] Handy JM, Soni N. Physiological effects of hyperchloraemia and acidosis. Br J Anaesth. 2008 Aug;101(2):141-50. doi: 10.1093/bja/aen148. Epub 2008 Jun 4. PMID 18534973
- [Background] Kiely DG, Cargill RI, Lipworth BJ. Effects of hypercapnia on hemodynamic, inotropic, lusitropic, and electrophysiologic indices in humans. Chest. 1996 May;109(5):1215-21. doi: 10.1378/chest.109.5.1215. PMID 8625670
- [Background] Onwochei D, El-Boghdadly K, Oakley R, Ahmad I. Intra-oral ignition of monopolar diathermy during transnasal humidified rapid-insufflation ventilatory exchange (THRIVE). Anaesthesia. 2017 Jun;72(6):781-783. doi: 10.1111/anae.13873. Epub 2017 Mar 20. PMID 28321836
- [Background] Akhtar N, Ansar F, Baig MS, Abbas A. Airway fires during surgery: Management and prevention. J Anaesthesiol Clin Pharmacol. 2016 Jan-Mar;32(1):109-11. doi: 10.4103/0970-9185.175710. PMID 27006554
- [Derived] Kuo YT, Chang TS, Tsai CC, Chang HC, Chia YY. Optimizing nonintubated laryngeal microsurgery: The effectiveness and safety of superior laryngeal nerve block with high-flow nasal oxygen-A prospective cohort study. J Chin Med Assoc. 2024 Mar 1;87(3):334-339. doi: 10.1097/JCMA.0000000000001057. Epub 2024 Jan 30. PMID 38305707